CLINICAL TRIAL: NCT02755883
Title: Strides For Life I: A Randomized Controlled Trial of Induction of Positive Affect to Increase Physical Activity in Early Stage Lung Cancer Survivors
Brief Title: Strides for Life I: Increasing Physical Activity in Stage 1 Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Lung Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1510016644
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
Keywords: Physical activity; non-small lung cancer; positive affect
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical activity plus positive affect (Experimental): Subjects will be randomized to a physical activity goal and the positive affect component
  Interventions: Behavioral: Physical activity plus positive affect
- Physical activity plus education (Active Comparator): Subjects will be randomized to a physical activity goal and education
  Interventions: Behavioral: Physical activity plus education

INTERVENTIONS:
Behavioral: Physical activity plus positive affect — Subjects will be randomized to a physical activity goal and will receive the positive affect component.
  Arms: Physical activity plus positive affect
Behavioral: Physical activity plus education — Subjects will be randomized to a physical activity goal and will receive the educational component.
  Arms: Physical activity plus education

SUMMARY:
This randomized controlled trial will evaluate, among 54 stage early stage lung cancer patients, whether a behavioral intervention versus an educational Control group results in improved function at 6-months.

DETAILED DESCRIPTION:
This is a two arm randomized controlled trial that will evaluate, among 54 stage 1 non-small cell lung cancer patients, whether induction of positive affect vs. an educational Control group, results in improved function as assessed by the 6-minute Walk Test. Our primary outcome will be a within-patient change in the 6-Minute Walk Test at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer (Stage 1)

Exclusion Criteria:

1. Cognitive impairment
2. Inability to walk
3. < 12 month anticipated survival
4. enrollment in other behavioral programs
5. lack of medical approval to participate
6. substance/alcohol dependence or participation in a substance abuse treatment program within 12 months
7. major psychiatric illness.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Kilocalories/week assessed by 6-minute walk test | 1 month to 6 months

SECONDARY OUTCOMES:
Forced expiratory volume (FEV1) | 1 month to 6 months
  Pulmonary function test
Functional Assessment of Cancer Therapy- Lung (FACT-L14) | 1 month to 6 months
  Disease-specific quality of life
Activity expenditure (assessed by the Fit Bit Zip accelerometer) | 1 month to 6 months
Maximal Oxygen Consumption (VO2 max) | 1 month to 6 months
  Pulmonary function test

CONTACTS AND LOCATIONS:
Overall Officials: Janey Peterson, EdD, MS, RN, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided